CLINICAL TRIAL: NCT02818881
Title: Differences in Energy Expenditure of Two Commonly Used Yoga Protocols
Brief Title: Electromyography and Yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20140550
Record Dates: First submitted 2016-06-23; First posted 2016-06-30 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Yoga
Keywords: aerobic; muscle activity; energy expenditure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-speed then low-speed yoga (Experimental): Subjects received a single session of High-speed yoga and within one week a single session of Low-speed yoga
  Interventions: Other: High-speed yoga; Other: Low-speed yoga
- Low-speed then high-speed yoga (Experimental): Subjects received a single session of Low-speed yoga and within one week a single session of High-speed yoga
  Interventions: Other: High-speed yoga; Other: Low-speed yoga

INTERVENTIONS:
Other: High-speed yoga
Other: Low-speed yoga

SUMMARY:
This study examined the muscle activity, movement patterns, and oxygen consumption during a series of yoga poses with slow and rapid transitions.

ELIGIBILITY:
Inclusion Criteria:

* Have at least 1 year of yoga experience;
* Practice a minimum of twice per week (app 2 hours or more);
* Demonstrate good form in the poses (asanas) making up the Sun A and Sun B sequences;

Exclusion Criteria:

* If they have any uncontrolled neuromuscular, orthopedic or cardiovascular disease;
* If they have been advised by their physicians that they should not exercise;
* If they cannot complete three cycles each of the Sun A and B sequence in good form.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Comparison of energy expenditures for high-speed and low-speed yoga | Day 3
  We measured calories for all subjects across both conditions

SECONDARY OUTCOMES:
Comparison of muscle activities for high-speed and low-speed yoga | Day 3
  We measured muscle activities for all subjects across both conditions
Comparison of oxygen utilization for high-speed and low-speed yoga | Day 2
  We measured oxygen consumption for all subjects across both conditions

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Max Orovitz Laboratory, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No